CLINICAL TRIAL: NCT00283504
Title: A Description of Inflammatory Cell Types in Moderate to Severe Pediatric Asthma: Eosinophilic and Non Eosinophilic Sputum Markers While on Anti-IgE Therapy (Xolair)
Brief Title: A Description of Inflammatory Cell Types In Moderate to Severe Pediatric Asthma: Eosinophilic and Non Eosinophilic Sputum Markers While on Anti-IgE Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of The King's Daughters (Other)
Collaborators: Novartis (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, MARIPAZ B. MORALES MD, MD, Children's Hospital of The King's Daughters
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB# 05-08-EX-0247
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: ALLERGIC ASTHMA
MeSH Terms: interventions — Omalizumab

ARMS (1):
- all patients received Xolair/active drug (Experimental): One arm:active drug
  Interventions: Drug: ANTI-IGE THERAPY (XOLAIR)

INTERVENTIONS:
Drug: ANTI-IGE THERAPY (XOLAIR) — Xolair dosing is based on body weight and baseline serum total IgE concentration(0.016 x kg body weight x IgE levels), with a maximum dose per 4 weeks of 750mg.Depending on their weight and IgE levels, patients get their Xolair shots every 2 or every 4 weeks.

SUMMARY:
The researcher proposes to assess levels of sputum inflammatory markers (eosinophils, eosinophil cationic protein (ECP), neutrophils IL-8) before and while on anti-IgE therapy in a pediatric population of moderate to severe asthmatics who have ongoing persistent asthma symptoms despite on moderate to high doses of inhaled corticosteroids (ICS).

Associations will be assessed between the types of sputum inflammatory markers and the patient's atopic status and level of asthma control as indicated by the following measures:

1. pulmonary function test (PFT)
2. asthma symptoms based on the Asthma Control Test (ACT)

DETAILED DESCRIPTION:
Objectives:

Primary: Describe inflammatory cell types in study patients and compare changes in inflammatory cell patterns before and during anti-IgE therapy.

Secondary:Describe patterns of sputum eosinophilia and neutrophilia in relation to asthma symptom improvement based on ACT and PFT

Hypotheses:

Differences in inflammatory response after the addition of anti-IgE therapy can be described in neutrophilic, eosinophilic and neutrophilic/eosinophilic asthmatics.

Neutrophilic asthmatics patients will fail to respond when placed on anti-IgE while eosinophilic asthmatics will respond well.

Sputum inflammatory markers are sensitive markers of inflammation and can predict response to new asthma treatment modalities such as anti-IgE therapy.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe allergic asthma, uncontrolled on conventional therapy

Exclusion Criteria:

* History of systemic illness, currently on other immune modulators like immunotherapy, IVIg
* Pregnancy
* IgE level >1300

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MARIPAZ B MORALES, MD, Principal Investigator — CHILDREN'S HOSPITAL OF KING'S DAUGHTERS/EASTERN VIRGINIA MEDICAL SCHOOL

RESULTS

PARTICIPANT FLOW:
Groups:
- Eosinophilic Phenotype; Non Eosinophilic Phenotype: participants received Xolair per standard clinical practice
Period: Overall Study
Arm/Group | Eosinophilic Phenotype | Non Eosinophilic Phenotype
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eosinophilic Phenotype | Non Eosinophilic Phenotype | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 6 | 13
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 13
number of participants with eosinophilic or non eosinophilic (neutrophilic) sputum [Count of Participants; unit: Participants] — The category of eosinophilic patients were based on their sputum eosinophils of >2.5% of total cells. The non eosinophilic patients on the other hand have >50% of neutrophils and <2.5 % eosinophils in their total sputum cells.
  Participants
    eosinophilic sputum | 7 | 0 | 7
    neutrophilic sputum | 0 | 6 | 6
asthma severity [Count of Participants; unit: Participants]
  severe | 5 | 2 | 7
  moderate | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Change in Sputum Markers by End of Study
Description: sputum markers were classified as eosinophilic or non eosinophilic
Time Frame: 32 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Eosinophilic Phenotype; Non Eosinophilic Phenotype: participants received xolair per standard practice
Arm/Group | Eosinophilic Phenotype | Non Eosinophilic Phenotype
Number analyzed (Participants) | 7 | 6
Participants | 0 | 0

2. Secondary Outcome: Number of Participants With Response to Therapy Based on Clinical Parameters Such as ED Visits, Hospitalizations, Systemic Steroid Use and Symptom Control
Time Frame: 32 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Eosinophilic Phenotype | Non Eosinophilic Phenotype
Number analyzed (Participants) | 7 | 6
Participants | 7 | 6

3. Secondary Outcome: Number Participants for Whom Sputum Induction Was Safe
Description: safety was assessed by measuring FEV1 levels before and after sputum induction; induction was considered safe if FEV1 levels remained the same or improved
Time Frame: every 4 weeks up to 32 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Eosinophilic Phenotype | Non Eosinophilic Phenotype
Number analyzed (Participants) | 7 | 6
Participants | 7 | 6

ADVERSE EVENTS:
Arm/Group | Eosinophilic Phenotype | Non Eosinophilic Phenotype
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

LIMITATIONS AND CAVEATS:
Difficulty enrolling patients and therefore had a small study population, limiting the results of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No